CLINICAL TRIAL: NCT03251274
Title: The Effect of Eddy Current Function of Bath Machine on Sleep Quality in Nursing Home
Brief Title: Bath Machine on Sleep Quality in Nursing Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CMUH105-REC3-138
Record Dates: First submitted 2017-07-28; First posted 2017-08-16 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Sleep
Keywords: bath machine; sleep quality; nursing home; heart rate variability
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: machine bathing group traditional bathing group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- machine bathing group (Experimental): structured machine bathing for 20-min duration at evening.
  Interventions: Other: machine bathing
- traditional bathing group (Active Comparator): traditional bathing at evening.
  Interventions: Other: traditional bathing

INTERVENTIONS:
Other: machine bathing — machine bathing 20-min duration at evening
  Arms: machine bathing group
Other: traditional bathing — traditional bathing
  Arms: traditional bathing group

SUMMARY:
The study is divided into two stages, the purposes of the first stage are (1) to examine the feasibility and simplicity of the operation of bathtub machine for nurse aides; (2) to examine the safety and comfortability of the bathtub machine from the perspectives of the nurse aides. The purposes of the second stage are (1) to understand the experiences of nurse aides and the elderly with disability by using the bathtub machine(which has edde massage function); (2) to evaluate the effectiveness of using the bathtub machine on the sleep quality and body temperature in the elderly with disability.

DETAILED DESCRIPTION:
The trends of bath disability in elderly consistently increased and, enhance, the demand of helping bath for the elderly also increased in Taiwan. Bathing is an important item of activities of daily living for human. Bathing not only keeps the body clean but also makes body comfort. Some studies showed that taking hot (40-40.5°C) baths 1.5 - 2 hours before bedtime resulted in a significant increase slow wave sleep (SWS) in the early part of the sleep period and improving sleep continuity in older female insomniacs.

Nurse aides are one of important human resource for long-term care institution. In Taiwan, Chao et al. reported that nurse aides had long-term accumulating discomfort over neck, shoulders and lower back during helping disable residents to carry out activity daily life. However, the body discomfort in nurse aides significantly decreased by using auxiliary equipment during assisting the elderly to carry out activity daily life. Therefore, it is important to use auxiliary equipment to prevent injury during work for nurse aides.

This study is interested in applying edde massage bathtub to improve sleep quality for disable residents in long-term care institutions. The study is divided into two stages, first stage of the study is to train nurse aides to use the bathtub machine (which has edde massage function) and solicits the opinions of nurse aides about factors related to the accessibility and safety of bath-tub machine using focus group methods. The purposes of the first stage study are (1) to examine the feasibility and simplicity of the operation of bathtub machine for nurse aides; (2) to examine the safety and comfortability of the bathtub machine from the perspectives of the nurse aides.

Second stage of the study is to explore the experiences of nurse aides and disabled elderly by using the bathtub machine. The purposes of the second stage study are (1) to understand the experiences of nurse aides and the elderly with disability by using the bathtub machine(which has edde massage function); (2) to evaluate the effectiveness of using the bathtub machine on the sleep quality and body temperature in the elderly with disability.

ELIGIBILITY:
Inclusion Criteria:

* More than half a year in the institution
* 18 years of age (including) or above, with the help of bathing
* Be conscious, able to listen, speak Chinese

Exclusion Criteria:

* Acute illness
* Diabetes
* Peripheral blood vessels or neurological diseases
* Mental disorders
* Sleep apnea
* Long-term hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
sleep quality | the night after intervention
  Polysomnography, PSG

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Liang Lai, Principal Investigator — Taichung Hospital, Ministry of Health and Welfare
Locations (1):
- Taichung Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
participant's data of polysomnography and heart rate variability can be shared